CLINICAL TRIAL: NCT02635555
Title: The Effects of Height and Weight Adjusted Dose of Local Anesthetic Compared to Standard Dose for Spinal Anesthesia in Elective Cesarean Section
Brief Title: The Effects of Height and Weight Adjusted Dose of Local Anesthetic.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shalini Dhir, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 107445
Record Dates: First submitted 2015-12-10; First posted 2015-12-21 (Estimated); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Complications; Cesarean Section; Hypotension
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine; Ephedrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adjusted Spinal Dose (Experimental): Patients in this group receive height and weight adjusted dose for spinal anesthesia.During surgery, phenylephrine/ephedrine is given to maintain blood pressure as necessary.
  Episodes of hypotension will be treated with these vasopressors .
  Interventions: Drug: Phenylephrine
- Standard Spinal Dose (Active Comparator): Patients in this group receive a fixed standard dose for spinal anesthesia. During surgery, phenylephrine/ephedrine is given to maintain blood pressure as necessary.
  Episodes of hypotension will be treated with these vasopressors .
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Phenylephrine — 100 mcg of phenylephrine or 5 mg ephedrine given as deemed necessary for treating episodes of hypotension.
  Other Names: Ephedrine

SUMMARY:
At our centre a conventional dose of 12 mg of hyperbaric bupivacaine in combination with a short acting opioid fentanyl (to increase block density) and a long acting opioid morphine (to provide post-operative pain relief ) is used for spinal anesthesia for cesarean section.However, larger doses of local anesthetic drug when used in caesarean section commonly cause low blood pressure and requires drugs (vasopressors) to treat it. In our study the investigators will standardize the doses of both opioids (fentanyl/morphine) and adjust the dose of local anesthetic (bupivacaine) based on the patients height and weight .One of the obvious challenges anesthesiologists face is providing adequate anesthesia to the patient whilst minimizing harmful side effects. Our primary concern is the low blood pressure as an effect of the spinal anesthetic as it is harmful to both mother and the baby. The investigators propose that the extent of surgical anesthetic block, which is dependent on height and weight in our adjusted dose group, will provide adequate anesthesia for surgery and minimise maternal low blood pressure.

DETAILED DESCRIPTION:
Study design is prospective, randomized, double blind, placebo controlled.

Patients presenting for elective cesarean section under neuraxial block and meeting inclusion criteria will be randomized to two groups:

Group 1: Fixed dose group: Bupivacaine 12 mg, Fentanyl 15 mcg, Morphine 100 mcg Group 2: Height and weight adjusted bupivacaine dose, fentanyl 15 mcg, morphine 100 mcg Patients are fasted as per Canadian guidelines prior to the procedure. All patients have an IV cannula inserted,baseline vitals recorded and routine blood work checked prior to blockade. Routine monitoring (as per Canadian Anesthesia Society (CAS) guidelines) occur during and after the procedure. This includes pulse oximetry (SpO2), ECG and non-invasive blood pressure (NIBP). NIBP monitoring occurs every two minutes for the first 20 minutes post spinal and every 5 minutes thereafter. Oxygen via Hudson mask or nasal prongs is available if required.

Spinal anesthetic is performed with standard doses of drugs and the level of sensory block is tested with ice. Motor block is tested with Bromage scale just before prepping and draping. Once deemed adequate, surgery begins. During surgery, phenylephrine/ephedrine is given to maintain blood pressure as necessary. After surgery, patients are monitored in a recovery area until fit to be transferred to their rooms. If patient reports extreme discomfort or sharp pain during the surgery,conversion to general anesthetic is as per the discretion of the attending anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

ASA I and II patients aged 18-40 > 37 weeks gestation

* Scheduled for an elective c-section under spinal anesthetic
* Singleton pregnancy
* Patients height between 150-180cm and with a BMI of <35
* Subject understands the study and consents to participate

Exclusion Criteria:

Contraindication to neuraxial blockade

* Local anesthetic allergy
* Above or below our defined height and BMI criteria
* Emergency C-Section
* Complicated pregnancy including severe toxemia, pregnancy induced hypertension, and placenta previa

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Maternal hypotension needing vasopressors. | Until the end of surgery

SECONDARY OUTCOMES:
Time to adequate surgical anesthetic block | 24 hours after the surgery
incidence of nausea, vomiting, pruritus, and respiratory depression | 24 hours after the surgery
conversion to general anesthesia due to block failure | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Dhir, FRCPC, Principal Investigator — Western University
Locations (1):
- Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No